CLINICAL TRIAL: NCT01626248
Title: Analysis of Lymphocyte Cell Surface Adhesion Marker Expression in a Natalizumab Treated Population With Active Control Assessment
Brief Title: Analysis of Lymphocyte Cell Surface Adhesion Marker Expression in Natalizumab Population With Active Control
Status: Completed | Type: Observational
Sponsor: John F. Foley, MD (Other)
Collaborators: Biogen (Industry); Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, John F. Foley, MD, President, Sponsor-Investigator, Rocky Mountain MS Research Group, LLC
Organization: Rocky Mountain MS Research Group, LLC (Other)
Other Study IDs: 005-001-TY
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Multiple Sclerosis
Keywords: Immunological; biomarkers; observational; RRMS; Relapsing; Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Recurrence

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Group A TX Naive: Patient decided to start disease modifying treatment, either interferon beta-1a, glatiramer acetate or natalizumab. If interested and consented they would be assigned to Group A. Patient would have blood specimens taken up to 5 times over the next 19 months: Day 0; Day 28; Day 84: Day 336 and Day 508.
- Group B TY 4-12 doses: Patient is currently prescribed and is taking natalizumab, has 4 to 12 doses. If interested patient could be consented and assigned to Group B. Patients will have their blood drawn Day 0; and around the time of the patient's 18th dose.
- Group C 18 plus TY: Patient currently or close to being at 18 doses or 18 plus doses of natalizumab. If interested patient consented and assigned to Group C. Patient will have their blood drawn once: Day 0.
- Group D Other DMT 18 plus: Patient is close to or currently at 18 doses or more of interferon beta-1a or glatiramer acetate. If interested patient consented and assigned to Group D. Patient will have their blood drawn once: Day 0.
- Group E - Non-MS: 10 participants without Multiple Sclerosis or other immunological illness. If interested participants consented and assigned to Group E. Participants will have their blood drawn once: Day 0.

SUMMARY:
The purpose of the study is to research the association between receiving Tysabri® (natalizumab), interferon beta-1a, glatiramer acetate or not having any treatment for your MS and how it may or may not impact certain white blood cells and other immunological markers. This information may be useful in identifying risk factors in developing progressive multifocal leukoencephalopathy (PML). It does appear that the risk increases with the total number of natalizumab infusions. Patients who have not yet started a disease modifying therapy or who have been on one other than natalizumab are needed as controls to see how these biomarkers change.

Patients at various stages of natalizumab treatment as well as natalizumab naïve are needed to allow for analysis of the change in potential markers over time.

DETAILED DESCRIPTION:
Patients at various timepoints in their MS treatment or who are beginning certain MS treatments will be consented and have blood specimens collected to allow for an immunological comparison. The decision to treat with disease modifying therapies is made independently from this observational study.

Primary endpoint: To further understand the delineation of lymphocyte cell adhesion marker down regulation within a treatment naïve patient population and at various stages of treatment.

Secondary endpoint: To understand the correlation between natalizumab pharmacodynamics, pharmacokinetics and lymphocyte cell adhesion marker down regulation.

The results of various biomarkers and immunological testing (including CD62L, LFA-1, sCD62L, sLFA-1, sVCAM, VLA-4 saturation, IgG4, CBC with absolute differential) will be compared amongst the groups consented. The treatment naive group will be compared longitudinally.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
2. Aged 18 to 80 years old, inclusive, at the time of informed consent.
3. Patients with a relapsing form of Multiple Sclerosis as determined by the treating or back-up neurologist per chart review.
4. If getting natalizumab or scheduled to commence natalizumab infusion the patient must be enrolled in the TOUCH Prescribing Program and who is not expected to discontinue Tysabri® therapy prior to completion of the requirements of this study or must be currently prescribed and using interferon beta 1a or glatiramer acetate injections for 18 months; or, naïve to natalizumab, interferon beta 1a or glatiramer acetate and beginning treatment after consent.
5. Patients screened for Group A must be completely naïve to natalizumab, patients beginning interferon beta-1a or glatiramer acetate must also be naïve to natalizumab.
6. Patients screened for natalizumab naïve must have at least 30 days clear of other disease modifying therapies.
7. Patients must be free of known systemic bacterial or viral infections.
8. No fever over 99.5 degrees Fahrenheit in the last two weeks or at Baseline or prior to any scheduled specimen collection.
9. No herpes zoster outbreaks within the last 30 days.
10. No methylprednisolone sodium succinate infusion (solumedrol) or corticosteroid use within the last 30 days.
11. Must weigh between 44 and 190 kg, inclusive.

Exclusion Criteria:

1. Patient is unwilling or unable, in the opinion of the investigator, to comply with study instructions.
2. Patients experiencing a MS relapse or exacerbation which results in methylprednisolone sodium succinate infusion 30 days prior to Baseline
3. Patients with active, unknown infection etiology - if a patient is being treated for a known infection this would be allowed at the discretion of the Investigator, but if they present with signs of infection that has not been diagnosed they should be excluded.
4. Fever of 99.6 or higher within the last two weeks prior to any of the scheduled specimen collection (Baseline, 1 month, 3 month, 12 month or 18 month).
5. If patient has missed doses of their DMT as per the inclusion criteria.
6. No prior immunosuppressant use (e.g., mitoxantrone, azathioprine, methotrexate, cyclophosphamide, mycophenolate mofetil).
7. Specimen collection must occur Monday through Thursday.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Relapsing Remitting Multiple Sclerosis (RRMS) who are treated at Rocky Mountain Multiple Sclerosis Clinic, and who are currently undergoing disease modifying therapy, natalizumab, glatiramer acetate injections, interferon beta 1a, or who are beginning one of these disease modifying therapies.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Quantitative Assessment of CD62L in MS Patients on Immunomodulatory Agents | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: John F Foley, MD, Principal Investigator — Rocky Mountain MS Research Group, LLC
Locations (1):
- Rocky Mountain MS Clinic, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Berger T, Rubner P, Schautzer F, Egg R, Ulmer H, Mayringer I, Dilitz E, Deisenhammer F, Reindl M. Antimyelin antibodies as a predictor of clinically definite multiple sclerosis after a first demyelinating event. N Engl J Med. 2003 Jul 10;349(2):139-45. doi: 10.1056/NEJMoa022328. PMID 12853586
- [Background] Harris VK, Sadiq SA. Disease biomarkers in multiple sclerosis: potential for use in therapeutic decision making. Mol Diagn Ther. 2009;13(4):225-44. doi: 10.1007/BF03256329. PMID 19712003
- [Background] Rice GP, Hartung HP, Calabresi PA. Anti-alpha4 integrin therapy for multiple sclerosis: mechanisms and rationale. Neurology. 2005 Apr 26;64(8):1336-42. doi: 10.1212/01.WNL.0000158329.30470.D0. PMID 15851719
- [Background] Shimada Y, Hasegawa M, Takehara K, Sato S. Elevated serum L-selectin levels and decreased L-selectin expression on CD8(+) lymphocytes in systemic sclerosis. Clin Exp Immunol. 2001 Jun;124(3):474-9. doi: 10.1046/j.1365-2249.2001.01514.x. PMID 11472411